CLINICAL TRIAL: NCT07366905
Title: Clinical Observation of Bupivacaine Liposome for Lower Extremity Femoral Nerve Block
Brief Title: Clinical Observation of Bupivacaine Liposome for Lower Extremity Nerve Block
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hainan Medical College (Other)
Collaborators: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Principal Investigator, Xin Chen, Associate researcher, Hainan Medical College
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUMU2H-DCOEOP-CN-2025; No.823RC592 (Other Grant/Funding Number: Hainan Provincial Natural Science Foundation of China)
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Patients Eligible for Elective Lower Extremity Femoral Nerve Surgery; Knee Arthroscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasound-guided femoral nerve block with liposomal bupivacaine (Experimental): Participants receive ultrasound-guided femoral nerve block with liposomal bupivacaine administered at varying concentrations using a modified up-and-down sequential dose-finding design. Sensory and motor block responses are assessed 30 minutes after block placement to estimate EC50 and EC95.
  Interventions: Drug: Liposomal bupivacaine, 266mg

INTERVENTIONS:
Drug: Liposomal bupivacaine, 266mg — Liposomal bupivacaine administered for ultrasound-guided femoral nerve block at varying concentrations using a modified up-and-down sequential dose-finding design.

SUMMARY:
This prospective, sequential dose-finding clinical observational study aims to estimate the median effective concentration (EC50) and the 95% effective concentration (EC95) of liposomal bupivacaine for ultrasound-guided femoral nerve block. Sensory and motor block endpoints are evaluated separately at 30 minutes after block placement using a modified up-and-down (sequential allocation) design, with trial termination after eight reversal points.

DETAILED DESCRIPTION:
This prospective clinical observational, sequential dose-finding study is designed to determine the effective concentrations of liposomal bupivacaine for ultrasound-guided femoral nerve block in patients undergoing lower limb surgery or related procedures.

All patients receive ultrasound-guided femoral nerve block performed by an experienced anesthesiologist using a standardized technique. A fixed injection volume of liposomal bupivacaine is administered, while the drug concentration is adjusted according to a modified up-and-down sequential method. The concentration for each subsequent participant is determined based on the response of the preceding participant. Following a positive response, the concentration is decreased; following a negative response, the concentration is increased by a pre-specified step size. The study is terminated after eight reversal points (crossovers) are observed.

To independently characterize sensory and motor block dose-response relationships, participants are allocated into two endpoint-specific observation groups:

Sensory block group

Sensory function in the femoral nerve distribution is assessed 30 minutes after block placement using standardized sensory testing. Complete loss of sensation at 30 minutes is defined as a positive response, while preserved sensation is defined as a negative response.

Motor block group

Motor function of the quadriceps muscle is evaluated 30 minutes after block placement using a standardized motor strength assessment. Complete loss of quadriceps muscle strength or paralysis at 30 minutes is defined as a positive response, while preservation of motor function is defined as a negative response.

The primary objective of this study is to estimate the EC50 and EC95 of liposomal bupivacaine for:

femoral nerve sensory blockade, and

femoral nerve motor blockade,

based on sequential allocation data and appropriate dose-response modeling.

Secondary objectives include describing the differential sensory-motor block profile of liposomal bupivacaine and evaluating its clinical feasibility and safety for femoral nerve block applications. All patients are monitored for block-related adverse events, including signs of local anesthetic systemic toxicity, nerve injury, and other complications throughout the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years
* Scheduled for elective unilateral lower limb surgery
* Unilateral ultrasound-guided femoral nerve block clinically indicated as part of routine perioperative anesthesia and analgesia management
* Ability to clearly distinguish between the blocked (operated) limb and the contralateral (non-blocked) limb for sensory and pain assessments
* Ability to understand the study procedures and provide written informed consent
* Ability to cooperate with sensory and motor assessments, including visual analog scale (VAS) scoring and quadriceps muscle strength testing

Exclusion Criteria:

* Known allergy or hypersensitivity to bupivacaine, amide-type local anesthetics, or any component of liposomal bupivacaine
* Infection at or near the planned injection site
* Coagulopathy or clinically significant bleeding disorder, or anticoagulant/antiplatelet therapy incompatible with peripheral nerve block
* Pre-existing neurological deficits, neuropathy, or motor weakness affecting either lower limb that could interfere with sensory or motor assessments
* Severe hepatic dysfunction or other conditions that increase the risk of local anesthetic systemic toxicity
* Pregnancy or breastfeeding
* Emergency surgery
* Inability to complete study assessments or comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
EC50 and EC95 for femoral nerve sensory block | 30 minutes after femoral nerve block placement
  The median effective concentration (EC50) and the 95% effective concentration (EC95) of liposomal bupivacaine for ultrasound-guided femoral nerve sensory blockade are estimated using a modified up-and-down sequential dose-finding design.
  Sensory block is assessed 30 minutes after block placement in the femoral nerve distribution on the blocked side, including the anterior thigh (anterior femoral cutaneous nerve territory) and the medial aspect of the lower leg (saphenous nerve territory). Sensory testing is performed using pinprick testing and/or cold stimulation with an ether-soaked cotton swab, with the contralateral non-blocked limb used as an internal control.
  Sensory block is graded as follows: 0 = no block (sensation identical to the non-blocked limb); 1 = partial block (reduced sensation); 2 = complete block (absence of pain sensation). A positive sensory response is defined as a sensory block score of 2.
EC50 and EC95 for femoral nerve motor block | 30 minutes after femoral nerve block placement
  The median effective concentration (EC50) and the 95% effective concentration (EC95) of liposomal bupivacaine for ultrasound-guided femoral nerve motor blockade, estimated using a modified up-and-down sequential dose-finding design.
  Motor function is evaluated immediately after sensory assessment by assessing quadriceps muscle strength. Patients are instructed to perform a straight leg raise in the supine position or actively extend the knee. Muscle strength is graded using the Medical Research Council (MRC) scale (0-5).
  Motor function preservation is defined as an MRC score ≥4. A positive motor response (motor block) is defined as an MRC score ≤3, indicating clinically significant weakness or paralysis.

SECONDARY OUTCOMES:
Postoperative pain intensity assessed by VAS | 2, 6, 12, 24, and 48 hours postoperatively
  Postoperative pain intensity is assessed using the Visual Analog Scale (VAS, 0-10, where 0 indicates no pain and 10 indicates the worst imaginable pain). VAS scores are recorded separately for the operated (blocked) limb and the contralateral (non-blocked) limb. Pain assessments are performed at 2, 6, 12, 24, and 48 hours after surgery to evaluate postoperative pain progression and potential differences between limbs following femoral nerve block with liposomal bupivacaine.
Postoperative movement-evoked pain assessed by VAS | Postoperative day 1 and day 2
  Movement-evoked pain is assessed using the Visual Analog Scale (VAS, 0-10). VAS scores are recorded during active movement of the operated limb on postoperative day 1 and postoperative day 2 to evaluate pain associated with mobilization following femoral nerve block.
Quadriceps muscle strength after surgery | Postoperative day 1 and day 2
  Quadriceps muscle strength on the operated side is evaluated using the Medical Research Council (MRC) muscle strength scale (0-5). Assessments are performed on postoperative day 1 and postoperative day 2 to evaluate recovery of motor function following femoral nerve block.
Length of hospital stay | From the date of surgery until hospital discharge, assessed up to 30 days postoperatively.
  Length of hospital stay is defined as the number of days from the date of surgery to the date of hospital discharge.
Time to first ambulation after surgery | From the end of surgery until the first out-of-bed ambulation, assessed up to 72 hours postoperatively.
  Time to first ambulation is defined as the time interval from the end of surgery to the patient's first out-of-bed ambulation with or without assistance.
Intraoperative heart rate | From skin incision to the end of surgery, assessed continuously during the intraoperative period.
  Intraoperative heart rate is continuously monitored and recorded during surgery to assess intraoperative physiological stability.
Intraoperative mean arterial pressure | From skin incision to the end of surgery, assessed continuously during the intraoperative period.
  Intraoperative mean arterial pressure is continuously monitored and recorded during surgery to assess intraoperative hemodynamic stability.

OTHER OUTCOMES:
Adverse events related to femoral nerve block | From femoral nerve block placement until hospital discharge, assessed up to 30 days postoperatively.
  Adverse events potentially related to ultrasound-guided femoral nerve block or liposomal bupivacaine administration are monitored and recorded. These include, but are not limited to, local anesthetic systemic toxicity, nerve injury, infection, hematoma, and other block-related or drug-related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,the Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No